CLINICAL TRIAL: NCT01591083
Title: The Studies of the Pathophysiologic Mechanisms of Poor Ulcer Healing & Clinical Improvement to the High Ulcer Rebleeding Rate for Patients With Comorbid Illnesses
Brief Title: The Efficacy of Double Doses of Oral Esomeprazole in Preventing Rebleeding for Patients With Bleeding Peptic Ulcers
Acronym: DDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ER-100-008
Record Dates: First submitted 2012-05-02; First posted 2012-05-03 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Peptic Ulcer Bleeding
Keywords: Peptic ulcer rebleeding, double dose of esomeprazole
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Double oral dose (Active Comparator): Each enrolled patient receives an 80 mg loading dose of intravenous esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden) immediately after hemostasis was achieved spontaneously or by gastroscopy. Patients then received a 3-day continuous high dose (8 mg per hour) of esomeprazole infusion. Then, patients receive 40 mg oral esomeprazole twice daily for 11 days and followed by 40 mg once daily for 14 days.
  Interventions: Drug: esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden)
- Regular oral dose (Active Comparator): Each enrolled patient receives an 80 mg loading dose of intravenous esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden) immediately after hemostasis was achieved spontaneously or by gastroscopy. Patients then received a 3-day continuous high dose (8 mg per hour) of esomeprazole infusion. Then, patients receive 40 mg oral esomeprazole once daily for 25 days.
  Interventions: Drug: esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden)
- Control group (Active Comparator): Each enrolled patient receives an 80 mg loading dose of intravenous esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden) immediately after hemostasis was achieved spontaneously or by gastroscopy. Patients then received a 3-day continuous high dose (8 mg per hour) of esomeprazole infusion. Then, patients receive 40 mg oral esomeprazole once daily for 25 days.
  Interventions: Drug: esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden)

INTERVENTIONS:
Drug: esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden) — Each enrolled patient receives an 80 mg loading dose of intravenous esomeprazole (Nexium®, AstraZeneca AB, Södertälje, Sweden) immediately after hemostasis was achieved spontaneously or by gastroscopy. Patients then received a 3-day continuous high dose (8 mg per hour) of esomeprazole infusion. Then, patients with Rockall score >=6 are randomized into the double oral dose group and the regular oral dose group. Patients with Rockall score <6 are assigned to the control group.
  In the double oral dose group, patients receive 40 mg oral esomeprazole twice daily for 11 days and followed by 40 mg once daily for 14 days. In the other two groups, patients receive 40 mg oral esomeprazole 40 mg once daily for 25 days.
  Other Names: Nexium

SUMMARY:
Patients with comorbidities have an increased risk of ulcer re-bleeding, especially within the 14 days after first bleeding event. Three-day high dose esomeprazole infusion can prevent peptic ulcer rebleeding after endoscopic therapy. However, the optimal dose of oral esomeprazole is uncertain, especially for high risky patients. This study is to test whether a double dose of oral esomprazole could reduce peptic ulcer rebleeding for patients with Rockall score ≥ 6. Additionally, the second aim of this prospective study was to identify the selection criteria to predict poor fading and residual major stigmata of recent hemorrhage (SRH) or early recurrent bleeding after successful endoscopic hemostasis and high-dose PPI infusion.

DETAILED DESCRIPTION:
Peptic ulcer bleeding is a common and lethal disease, and the recurrent bleeding is an independent risk factor leading to the mortality. The recurrent bleeding of peptic ulcers is related to the presence of the stigmata of recent hemorrhage (SRH). The fading time of SRH is around 3 to 6 days, therefore, the recurrent bleeding develops within 2-3 days after first bleeding episode. The aim of acute treatment of peptic ulcer bleeding is to reduce recurrent bleeding by using anti-secretory drugs. Accordingly, the common duration of omeprazole infusion is applied as 3 days after the endoscopic therapy. Moreover, recurrent bleeding is also positively linked with the presence of co-morbidities. In general, patients with underlying medical co-morbidities have increased rates of recurrent bleeding and longer duration in risk of recurrent bleeding than those without co-morbidity.

Nonetheless, even with continuous infusion of omeprazole for 3 days, recurrent bleeding rates remain high in certain patients such as those with the presence of underlying medical co-morbidities. Moreover, the duration of peptic ulcer recurrent bleeding is elongated up to the 14th day after the first bleeding episode in patients with co-morbidities. To prevent recurrent bleeding in such high risk patients, we showed therapeutic benefit for the prolonged course of 7-day low-dose intravenous omeprazole, which exerts better recurrent bleeding control than just 3-day high-dose infusion.

The intragastric 24-h median pH is 4.9 in patients with oral 40 mg omeprazole once daily, which is significantly higher than baseline pH in healthy subjects. However, gastric acid secretion is not suppressed completely during 24 hours with oral omeprazole 40 mg once daily. Several studies have shown that oral high-dose PPI is equally effective in raising the intragastric pH more than 6 and reducing recurrent bleeding as the intravenous route.

Hence, this study aims to test whether a higher dose of oral esomeprazole, which is more effective in maintaining favorable intragastric pH, could effectively reduce ulcer rebleeding in patients with comorbidities. This data will show the originality and clinical importance of a higher dose of oral esomeprazole for such high-risk patients with comorbidities with peptic ulcer bleeding.

Additionally, endoscopic treatment plus a 3-day intravenous proton pump inhibitor infusion is the standard protocol for treatment of peptic ulcer bleeding. Moreover, several studies have shown that PPI treatment prior to endoscopy could decrease the presentation of SRH and the need of endoscopic hemostasis. However, there are insufficient data to validate the efficacy of such standard treatment to fade the SRH. Therefore, several studies looked at the efficacy of routine second-look endoscopy, defined as scheduled repeat endoscopy after primary endoscopic hemostasis in patients at high risk of rebleeding. However, the role of second-look endoscopy and the selection criteria for patients who require second-look endoscopy remain uncertain. There is a pressing need to elucidate the role of second-look endoscopy in patients with peptic ulcer bleeding after high-dose PPI infusion.

Hence, the second aim of this prospective study is to identify the selection criteria to predict poor fading and residual major SRH or early recurrent bleeding after successful endoscopic hemostasis and high-dose PPI infusion. This data will show the originality and clinical importance to identify the risk factors to predict poor fading of SRH after current standard treatment and the patients who are indicated to receive second-look endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received gastroscopy for melena, hematochezia, or hematemesis in whom bleeding peptic ulcers with major stigmata of recent hemorrhage are detected are consecutively enrolled. All of these major SRH are treated by local injection of diluted epinephrine 1:10000 with or without combined therapy with a heater probe, argon plasma coagulation, band ligation, or hemoclip therapy.

Exclusion Criteria:

* Patients are excluded if they had tumor bleeding or ulcer bleeding due to mechanical factors (i.e., gastrostomy tube induction), warfarin use, failure to establish hemostasis under gastroscopy, or hypersensitivity to esomeprazole or any component of the formulation.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
recurrent bleeding | within 28 days after the first bleeding event

SECONDARY OUTCOMES:
the length of hospitalization | within 28 days after the first bleeidng event
the amount of blood transfusion | within 28 days after the first bleeding event
major events such as surgery or transarterial embolization | within 28 days after the first bleeding event
the fading rate of major stigmata of recent hemorrhage | within 3 days after the first bleeding event
  At the primary gastroscopy, the adherent clot is vigorously washed away with water jet. All of the stigmata of recent hemorrhage (SRH) are treated by one or a combination of endoscopic therapies. The success of endoscopic hemostasis is defined as cessation of bleeding together with achievement of cavitation at the vessel after application of the heater probe.
  Second-look endoscopy is scheduled 48-72 hours after successful primary endoscopic hemostasis and intravenous high-dose proton pump inhibitor infusion. For each patient with either suspected or active recurrent bleeding, emergent endoscopy is conducted earlier before the schedule to confirm and treat peptic ulcer recurrent bleeding.
  Multiple logistic regression analysis is applied to assess the independent risk factors related to residual major stigmata or early recurrent bleeding of peptic ulcers.
mortality | within 28 days and 120 days after the first bleeding event

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Shyang Sheu, MD, Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan

REFERENCES:
- [Derived] Yang EH, Wu CT, Kuo HY, Chen WY, Sheu BS, Cheng HC. The recurrent bleeding risk of a Forrest IIc lesion at the second-look endoscopy can be indicated by high Rockall scores >/= 6. Surg Endosc. 2020 Apr;34(4):1592-1601. doi: 10.1007/s00464-019-06919-3. Epub 2019 Jun 20. PMID 31222633
- [Derived] Cheng HC, Yang EH, Wu CT, Wang WL, Chen PJ, Lin MY, Sheu BS. Hypoalbuminemia is a predictor of mortality and rebleeding in peptic ulcer bleeding under proton pump inhibitor use. J Formos Med Assoc. 2018 Apr;117(4):316-325. doi: 10.1016/j.jfma.2017.07.006. Epub 2017 Jul 24. PMID 28751088
- [Derived] Cheng HC, Wu CT, Chang WL, Cheng WC, Chen WY, Sheu BS. Double oral esomeprazole after a 3-day intravenous esomeprazole infusion reduces recurrent peptic ulcer bleeding in high-risk patients: a randomised controlled study. Gut. 2014 Dec;63(12):1864-72. doi: 10.1136/gutjnl-2013-306531. Epub 2014 Mar 21. PMID 24658598